CLINICAL TRIAL: NCT01715272
Title: A Clinical Investigation to Demonstrate the Performance of a New Enema (TF037) in Distal Bowel Cleansing Compared With Fleet Enema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NER1008-01/2012 (DBC)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy
MeSH Terms: interventions — sodium phosphate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fleet enema (Active Comparator): This group will receive Fleet enema as their treatment
  Interventions: Drug: Fleet enema
- TF037 (Experimental): This group will receive TF037 as their treatment
  Interventions: Device: TF037

INTERVENTIONS:
Device: TF037
  Arms: TF037
Drug: Fleet enema
  Arms: Fleet enema

SUMMARY:
This study is designed to assess the difference between the performance of a new enema (TF037) against Fleet enema in distal bowel cleansing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects [as determined by medical history, physical examination, laboratory test values, vital signs and 12-lead electrocardiograms (ECGs) at screening] aged 18 to 60 years.
* Non-smokers from 3 months before enema administration and for the duration of the clinical investigation.
* Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2.
* Must voluntarily provide written informed consent to participate in the clinical investigation.
* Must understand the purposes and risks of the clinical investigation and agree to follow the restrictions and schedule of procedures as defined in the clinical investigation plan, and as confirmed during the informed consent process.
* Female subjects must be postmenopausal (for at least one year and confirmed by a serum follicle stimulating hormone (FSH) test at screening), surgically sterile, practising true sexual abstinence or must use an effective method of contraception.
* Female subjects of child-bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in of each period.
* The subject's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical investigation.
* Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).

Exclusion Criteria:

* Subjects with a history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
* Subjects with a history or presence of organic or functional gastrointestinal conditions (e.g. chronic constipation, irritable bowel syndrome, inflammatory bowel disease).
* Subjects with a clinically relevant history or presence of abnormal gastrointestinal motility.
* Subjects with a significant history of hereditary bowel disorders.
* Subjects with abnormal findings on the digital rectal examination performed at screening.
* Use of laxatives or motility altering drugs in the 3 months preceding enema administration.
* Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 14 days prior to enema administration (or within 5 half lives if longer), with the exception of Investigator-approved hormonal contraceptives, hormone replacement therapy (HRT) and occasional paracetamol, aspirin or ibuprofen.
* Participation in a clinical drug study during the 30 days preceding enema administration in this clinical investigation.
* Donation of blood or blood products within 30 days prior to enema administration or during the clinical investigation, except as required for this clinical investigation
* Pregnant or lactating females.
* Any clinically significant illness within 28 days prior to enema administration.
* History or presence of any significant drug allergy, or a known allergy or contraindication to trisodium citrate, Fleet® enema or midazolam.
* Laboratory values at screening which are deemed to be clinically significant, unless agreed in advance by the Sponsor's Medical Representative and Principal Investigator.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Current or history of drug or alcohol abuse within the 12 months prior to enema administration, or a positive drugs of abuse test at screening or check-in.
* Consumption of alcoholic beverages within 24 hours of check-inor during confinement.
* Subjects who, in the opinion of the Investigator, are unsuitable for participation in the clinical investigation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Performance of TF037 in distal bowel cleansing compared to Fleet enema using the Harefield Cleansing scale | Between 1 to 3 hours following enema administration

SECONDARY OUTCOMES:
Stool output as measured by stool weight | up to 1 hour following enema administration
  To compare the stool output (as measured as stool weight) during the 1 hour period following enema administration for TF037 and Fleet enema
Safety and tolerability as assessed by use of a Visual Analogue scale (VAS) | 5 and 30 minutes following enema administration
  To assess the safety (including effects on water homeostasis) and tolerability of this medical device in its intended purpose
Stool output over time | 1 hour following enema administration
  To assess kinetics of bowel movements in relation to stool output over time

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Beboso, MD, Principal Investigator — BioKinetic Europe Ltd.
Locations (2):
- United Kingdom (2):
  - BioKinetic Europe Ltd, Belfast, Northern Ireland
  - BioKinetic Europe Ltd, Belfast